CLINICAL TRIAL: NCT06482086
Title: Precision Medicine Applied to Locally Advanced Thyroid Cancer Using Tumor-derived Organoids and In-vitro Sensitivity Testing: a Phase 2a, Single-center, Open-label, and Non-comparative Study
Brief Title: Efficacy of Organoid-Based Drug Screening to Guide Treatment for Locally Advanced Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Li Zhihui, Dean of the Thyroid Surgery Department, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202314711
Record Dates: First submitted 2024-06-15; First posted 2024-07-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Thyroid Gland Carcinoma
MeSH Terms: interventions — anlotinib; lenvatinib; Sorafenib; donafenib; Everolimus; apatinib; dabrafenib; trametinib; cabozantinib; vandetanib; entrectinib; pralsetinib; larotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organoid-guided targeted therapeutic group (Experimental): Patients who take the recommended drugs regularly based on sensitivity analysis.
  Interventions: Drug: Anlotinib; Drug: Lenvatinib; Drug: Sorafenib; Drug: Donafenib; Drug: Everolimus; Drug: Apatinib; Drug: Dabrafenib + Trametinib; Drug: Cabozantinib; Drug: Vandetanib; Drug: Entrectinib; Drug: Pralsetinib; Drug: Larotrectinib

INTERVENTIONS:
Drug: Anlotinib — 8/10/12 mg qd, po. Stop the medication for one week after taking it for two weeks.
Drug: Lenvatinib — 8/12 mg qd, po.
Drug: Sorafenib — 0.4 g bid, po.
Drug: Donafenib — 0.3 g bid, po.
Drug: Everolimus — 10 mg qd, po.
Drug: Apatinib — 500 mg qd, po.
Drug: Dabrafenib + Trametinib — Dabrafenib 150 mg bid, po+Trametinib 2 mg qd, po.
Drug: Cabozantinib — Cabozantinib 60mg qd, po.
Drug: Vandetanib — Vandetanib 300mg qd, po.
Drug: Entrectinib — Entrectinib 600mg qd，po.
Drug: Pralsetinib — 400mg qd, po.
Drug: Larotrectinib — 100mg qd，po

SUMMARY:
The current study aims to explore the potential advantages of anti-cancer therapy that is implemented based on drug sensitivity testing. This pertains to individuals with locally advanced thyroid cancer who have undergone conventional therapy in the past or unresectable patients .

DETAILED DESCRIPTION:
This research trial aims to determine the efficacy of organoid-guided targeted therapy for patients with locally advanced thyroid cancer. We will also investigate the variables affecting the effectiveness of targeted therapy for locally advanced thyroid cancer that is guided by organoids. Additionally, side effects related to the medication are also studied.

The following are the main questions that the trial seeks to address:

Can patients' tumor sizes be shrunk by taking medications that were found to be sensitive by organoid screening? Can patients' survival outcomes be improved by the medications that organoid screening found as sensitive? What aspects of the medications shown to be responsive by organoid screening are impacting their clinical efficacy? Is it possible for organoid-based drugs screening to guide treatment which lower surgical risk and make cancers that are now incurable into manageable ones? To ascertain the efficacy of the screened sensitive drugs in treating locally advanced thyroid cancer, researchers will measure the tumor size before and after taking the organoid-screened sensitive targeted drugs, assess the risk of radical resection, and document the survival outcomes of enrolled patients.

To further elucidate the parameters impacting the efficacy and prognosis, prognostic analysis based on clinical and pathological data, such as pathological type, gene mutation, age, tumor size, distant metastasis, and involvement of the trachea, esophagus, or major artery, will also be conducted.

The sample size for this study was determined based on the objective response rate (ORR) observed in our preliminary pilot study, which indicated an ORR of 22%. For papillary thyroid carcinoma (PTC), follicular thyroid carcinoma (FTC), and poorly differentiated thyroid carcinoma (PDTC), we aimed to detect a treatment effect with a minimum ORR of 12%, consistent with results from the previous multicenter, randomized, double-blind, placebo-controlled phase 3 trial (DECISION). For anaplastic thyroid carcinoma (ATC) and medullary thyroid carcinoma (MTC), we aimed to detect a treatment effect with a minimum ORR of 1%, considered the threshold for clinical efficacy.

To achieve a one-sided 95% confidence interval (α = 0.05), the Clopper-Pearson method was used to calculate the confidence interval for a proportion. This method ensured that the lower bound of the 95% confidence interval would exceed the minimum ORR (12% for PTC, FTC, and PDTC; 1% for ATC and MTC).

The calculation indicated that a total of 42 samples are needed for PTC, FTC, and PDTC, while 5 samples are required for both MTC and ATC.

Considering a 10% dropout rate and an 80% success rate for organoid drug sensitivity tests, a total of 59 samples are needed for PTC, FTC, and PDTC, while 7 samples are required for both MTC and ATC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult participants who have either been initially diagnosed with locally advanced thyroid cancer or have experienced persistent or recurrent thyroid cancer, including cervical nodal recurrence. Types of pathology include:

  1. Papillary thyroid carcinoma (PTC)
  2. Follicular thyroid carcinoma (FTC)
  3. Medullary thyroid carcinoma (MTC)
  4. Poorly differentiated thyroid carcinoma (PDTC)
  5. Anaplastic thyroid carcinoma (ATC)
* 2. Evidence of extrathyroidal extension and/or locally invasive disease and deemed at risk for R2 resection by treating team on clinical and/or fiberoptic examination and/or radiographic evaluation in the primary or recurrent setting. Evidence of "at risk for R2 resection" includes:

  1. Vocal cord paralysis by fiberoptic examination
  2. Extrathyroid and/or extranodal extension on CT or MRI, including tracheal and/or laryngeal cartilage invasion, esophageal involvement, and/or involvement of perithyroid muscles (e.g. strap, sternocleidomastoid, inferior constrictor muscles) or bone involvement
  3. Extension into the mediastinum with visceral and/or vascular involvement
  4. Involvement of the carotid artery or other major vessel by 180 degrees or more
  5. Other factors that make the participant to be "at risk for R2 resection" may be allowed, after discussion with the study's principal investigator.
* 3. There is at least one measurable lesion according to the Modified Response Evaluation Criteria in Solid Tumors (mRECIST).
* 4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
* 5. Normal organ and bone marrow function.
* 6. Adequate end-organ function (including bone marrow, coagulation, renal, liver and cardiac) 28 days prior to the study registration.
* 7. Ability to swallow pills.
* 8. Signed informed consent form.
* 9. Expected survival time of more than 2 months.

Exclusion Criteria:

* 1. Patients with contraindications specified in the drug instructions for the targeted drugs involved in the corresponding organoid drug sensitivity tests.
* 2. Patients with incomplete clinical data.
* 3. Patients with severe organ dysfunction, metabolic diseases, or other conditions significantly affecting survival.
* 4. Other active malignant disease requiring therapy.
* 5. Females who are pregnant or breastfeeding.
* 5. Patients without target lesions.
* 6. Patients deemed unsuitable for inclusion by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Every 8 weeks until progression up to 3 years
  ORR is defined as the percentage of patients who achieve a response, which can either be complete response (complete disappearance of lesions) or partial response (reduction in the sum of maximal tumor diameters by at least 30% or more)
Progress-free survival | Every 8 weeks until progression or death up to 3 years
  PFS is defined as the time from the administration of the first dose to first disease progression or death.
Overall R0/R1 resection rate | Up to 36 months.
  Defined as the proportion of patients who undergo R0/R1 resection among all patients.

SECONDARY OUTCOMES:
Overall Survival | Up to 36 months.
  OS is defined as the time from the administration of the first dose to death.
Change in Surgical complexity and morbidity score (SCMS) | Up to 36 months
  The Thyroid Neck Group Morbidity Complexity Scoring and MGH/MEE-MSK-MD Anderson (MMM) Surgical Morbidity Complexity Score (SMCS) are incorporated, specifying on scale with 5 levels of complexity and morbidity of the surgery [mild (level 0), moderate (level 1), severe (level 2), very severe (level 3), and unresectable (level 4)]. The surgical morbidity/complexity scores will be collected at enrollment, prior to surgery, and based on intraoperative findings.
  The change in SCMS will be reported as the median SCMS value. Determined by structures requiring resection, the score takes into account preoperatively radiographically defined structures judged to be requiring resection with surgical complexity of the given resection/potential for complications, and expected patient morbidity/change of function from the resection.
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v 5.0 | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhihui Li, Professor, Study Director — West China Hospital
Locations (1):
- West China hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo Z, Liu J, Zhang X, Ma Y, Wang Y, Li P, Huang R, Li Z; MDT of Advanced Thyroid Cancer of West China Hospital. Precision treatment guided by patient-derived organoids-based drug testing for locally advanced thyroid cancer: a single arm, phase 2 study. Endocrine. 2025 Jul;89(1):186-196. doi: 10.1007/s12020-025-04240-9. Epub 2025 Apr 30. PMID 40304938